CLINICAL TRIAL: NCT06674122
Title: The Efficacy of Enteral Vitamin D Supplementation at a Dose of 800 IU Compared to 400 IU in Preterm Infants With a Gestational Age of 28-34 Weeks Admitted to the Neonatal Care Unit
Brief Title: Efficacy of Higher Dose Enteral Vitamin D Supplementation in Preterm 28 - 34 Weeks of Gestational Age
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Rosalina Dewi Roeslani, Head of Neonatology Division, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VitD800vs400
Record Dates: First submitted 2024-11-01; First posted 2024-11-05 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Vitamin D Supplementation
Keywords: vitamin D supplementation in preterm

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400 IU (Active Comparator): Participants will receive enteral vitamin D supplementation of 400 IU/day for 28 days
  Interventions: Dietary Supplement: Enteral vitamin D supplementation of 400 IU/day
- 800 IU (Experimental): Participants will receive enteral vitamin D supplementation of 800 IU/day for 28 days
  Interventions: Dietary Supplement: Enteral vitamin D supplementation of 800 IU/day

INTERVENTIONS:
Dietary Supplement: Enteral vitamin D supplementation of 800 IU/day — Higher dose of enteral vitamin D supplementations (800 IU/day) are given for 28 days, and vitamin D status are examined before and after supplementation
  Arms: 800 IU
Dietary Supplement: Enteral vitamin D supplementation of 400 IU/day — Standard recommended dose of enteral vitamin D supplementations (400 IU/day) are given for 28 days, and vitamin D status are examined before and after supplementation
  Arms: 400 IU

SUMMARY:
The goal of this clinical trial is to learn about the effective dosage of enteral vitamin D supplementation in preterm infants with gestational age fom 28 to 34 weeks. The main questions it aims to answer is:

- Does higher dose of enteral vitamin D supplementation (800IU/day) increase vitamin D level better than standard recommended dose (400IU/day) to achieve sufficient level of vitamin D?

Participants will:

* Take the enteral vitamin D supplementation every fay for 28 days
* Have their blood level of vitamin D examined before and after supplementation for 28 days

DETAILED DESCRIPTION:
The study conducted in 2 hospitals in Jakarta region, RSCM and RSUD Koja. Preterm with 28 to 34 weeks of gestational age and fulfill the inclusion criteria will be enrolled in the study after parents signed the informed consent.

Blood sample will be collected to get the baseline of vitamin D serum. The study subject will be given enteral vitamin D supplementation for 28 days (4 weeks). The dosage of vitamin D is randomized with block randomized in sealed envelope.

Subjects then will be followed up to 28 days of supplementation. After 28 days of supplementation, the subjects' blood will be collected to get the vitamin D serum level. Data taken will be analyzed using IBM Statistical Product and Service Solutions (SPSS).

ELIGIBILITY:
Inclusion Criteria:

* neonates with gestational age 28-34 weeks
* tolerated enteral feedings more than 30ml/kg

Exclusion Criteria:

* infants with major congenital anomaly
* infants with gastrointestinal obstruction
* infants with congenital renal failure
* infants with cholestassis

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
25(OH)D level | From enrollment to the end of treatment at 4 weeks
  serum level of 25(OH)D

CONTACTS AND LOCATIONS:
Overall Officials: Rosalina D Roeslani, dr, SpA(K), Principal Investigator — FKUI RSCM
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Central Jakarta, Indonesia